CLINICAL TRIAL: NCT03263936
Title: Epigenetic Reprogramming in Relapse AML: A Phase 1 Study of Decitabine and Vorinostat Followed by Fludarabine, Cytarabine and G-CSF (FLAG) in Children and Young Adults With Relapsed/Refractory AML
Brief Title: Epigenetic Reprogramming in Relapse/Refractory AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2016-003
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2023-05

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Relapse; Myelogenous; Leukemia; Refractory; Acute; Pediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia | interventions — Decitabine; Vorinostat; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; fludarabine phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Other (Other): decitabine, vorinostat, fludarabine, high dose cytarabine, filgrastim (G-CSF)
  Interventions: Drug: Decitabine; Drug: Vorinostat; Drug: Filgrastim (G-CSF); Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Decitabine — Dose Level #0: 5 mg/m2 Dose Level #1: 7.5 mg/m2 Dose Level #2: 10 mg/m2 Dose Level #3: 15 mg/m2 Dose Level #4: 20 mg/m2 given IV over __ hour on days 1 through 5
  Other Names: Dacogen
Drug: Vorinostat — Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO.
  Other Names: Zolinza, SAHA, suberoylanilide acid
Drug: Filgrastim (G-CSF) — Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0)
  Other Names: G-CSF, neupogen
Drug: Fludarabine — 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF)
  Other Names: Fludara
Drug: Cytarabine — 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
  Other Names: Cytosine arabinoside, Ara-C, Cytosar

SUMMARY:
This is a pilot study using decitabine and vorinostat before and during chemotherapy with fludarabine, cytarabine and G-CSF (FLAG).

DETAILED DESCRIPTION:
Decitabine is a demethylating agent and vorinostat is a HDAC inhibitor. The use of demethylating agents and HDAC inhibitors in combination have been previously shown to have synergistic effects in altering neoplastic pathways of cancer cells and be well tolerated in human clinical studies. With the ability of decitabine and vorinostat to alter the abnormal cellular pathways of leukemic blasts and essentially turn off anti-apoptotic proteins, the leukemia cells have become primed for cytotoxic cell kill via chemotherapeutic agents. This study will ask the question as to whether or not the combination of decitabine and vorinostat followed by chemotherapy is feasible and whether it can positively impact outcome in patients with relapsed or refractory acute myelogenous leukemia.

ELIGIBILITY:
Inclusion Criteria:

- Patients must be ≥ 1 and ≤25 years of age.

Diagnosis: Patients with relapse or refractory AML must have measurable disease ( >M1 marrow)

* 1st or greater relapse, OR
* Failed to go into remission after 1st or greater relapse, OR
* Failed to go into remission from original diagnosis after 2 or more induction attempts

Eligibility for patients with an M1 marrow; defined as >0.1% by flow or molecular testing (e.g. PCR).

* must include two serial marrows (at least 1-week apart) demonstrating stable or rising minimal residual disease (MRD) (i.e. not declining).
* Patients may have CNS or other sites of extramedullary disease. No cranial irradiation is allowed during the protocol therapy.
* Patients with secondary AML are eligible.
* Patients with Down syndrome are eligible.
* Patients with DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Performance Level:

- Karnofsky >50% for patients >16 years of age and Lansky > 50% for patients ≤ 16 years of age (See Appendix II for Performance Scales)

Prior therapy - Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

1. Cytoreduction with hydroxyurea: hydroxyurea can be initiated and continued for up to 24 hours prior to the start of decitabine/vorinostat. It is recommended to use hydroxyurea in patients with significant leukocytosis (WBC >50,000/L) to control blast count before initiation of systemic protocol therapy.
2. Patients who relapsed while they are receiving cytotoxic therapy: at least 14 days must have elapsed since the completion of the cytotoxic therapy, except Intrathecal chemotherapy.

Hematopoietic stem cell transplant (HSCT):

- Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD) and are off all transplant immune suppression therapy for at least 7-days (e.g. steroids, cyclosporine, tacrolimus). Steroid therapy for non-GVHD and/or non-leukemia therapy is acceptable.

Hematopoietic growth factors:

- It must have been at least 7 days since the completion of therapy with GCSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta ®)

Biologic (anti-neoplastic agent):

-At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody (i.e. Gemtuzumab = 36 days)

Immunotherapy: At least 42 days after the completion of any time of immunotherapy, e.g. tumor vaccines or CAR T-cell therapy.

XRT: Cranio or craniospinal XRT is prohibited during protocol therapy. No washout period is necessary for radiation given to non-CNS chloromas; >90 days must have elapsed if prior TBI, cranio or craniospinal XRT.

Prior Demethylating and/or HDAC Inhibitor Therapy: Patients who have received prior DNMTi (e.g. decitabine) and/or HDACi (e.g. vorinostat) therapy are eligible to participate in this Phase 1 study. At least 7 days must have passed from prior DNMTi or HDACi as a washout period.

Renal and hepatic function: Patients must have adequate renal and hepatic functions as indicated by the following laboratory values:

A. Adequate renal function defined as: Patient must have a calculated creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2 OR a normal serum creatinine based on age/gender.

B. Adequate Liver Function Defined as: Direct bilirubin < 1.5 x upper limit of normal (ULN) for age or normal, AND alanine transaminase (ALT) < 5 x ULN for age. The hepatic requirements are waived for patients with known or suspected liver involvement by leukemia. This must be reviewed by and approved by the study chair or vice chair.

Adequate Cardiac Function Defined as: Shortening fraction of ≥ 27% by echocardiogram, OR ejection fraction of ≥ 50% by radionuclide angiogram (MUGA).

Reproductive Function A. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 1 week prior to enrollment.

B. Female patients with infants must agree not to breastfeed their infants while on this study.

C. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* No NG or G-Tube administration of Vorinostat is allowed. Capsule must be swallowed whole or given as oral suspension.
* They are currently receiving other investigational drugs.
* There is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* They have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* They have a known allergy to any of the drugs used in the study.
* Patients with DNA fragility syndromes are excluded (e.g. Fanconi Anemia, Bloom Syndrome)
* They are receiving valproic acid (VPA) therapy.
* Patients with Acute Promyelocytic Leukemia (APL, APML) are excluded
* Patients with documented active and uncontrolled infection at the time of study entry are not eligible

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (28):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - National Cancer Institute, Pediatric Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - CS Mott Children's Hospital, Ann Arbor, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - New York University Medical Center, New York, New York
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Cancer Center, Baylor, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - Sainte Justine University Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level #1: 7.5 mg/m2: Decitabine Dose Level #1: 7.5 mg/m2 given IV over 1 hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO on Days 1-5
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0) Days 5-12
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF) Days 6-10
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
- Dose Level #2: 10 mg/m2: Decitabine Dose Level #2: 10 mg/m2 given IV over 1 hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO on Days 1-5
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0) Days 5-12
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF) Days 6-10
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
- Dose Level #3: 15 mg/m2: Decitabine Dose Level #3: 15 mg/m2 given IV over 1 hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO on Days 1-5
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0) Days 5-12
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF) Days 6-10
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
Period: Overall Study
Arm/Group | Dose Level #1: 7.5 mg/m2 | Dose Level #2: 10 mg/m2 | Dose Level #3: 15 mg/m2
Started | 3 | 22 | 12
Completed | 3 | 20 | 12
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 (Decitabine = 7.5mg/m2): decitabine, vorinostat, fludarabine, high dose cytarabine, filgrastim (G-CSF)
  Decitabine Dose Level #1: 7.5 mg/m2
  given IV over __ hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO.
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0)
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF)
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
- Dose Level 2 (Decitabine 10mg/m2): decitabine, vorinostat, fludarabine, high dose cytarabine, filgrastim (G-CSF)
  Decitabine Dose Level #2: 10 mg/m2
  given IV over __ hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO.
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0)
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF)
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
- Dose Level 3 (Decitabine 15 mg/m2): decitabine, vorinostat, fludarabine, high dose cytarabine, filgrastim (G-CSF)
  Decitabine Dose Level #3: 15 mg/m2
  given IV over __ hour on days 1 through 5
  Vorinostat: Age <18: 180 mg/m2/day once daily PO. Age≥18: 200 mg twice daily PO.
  Filgrastim (G-CSF): Given on days 5 until evidence of ANC recovery (>500/µL)5µg/kg/dose IV or SQ (starting at hour 0)
  Fludarabine: 30 mg/m2/day IV over 30 minutes (starting at Hour 0 - Immediately after G-CSF)
  Cytarabine: 2000 mg/m2/day (Starting at Hour 0.5),IV over 3 hours, days 6-10
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (Decitabine = 7.5mg/m2) | Dose Level 2 (Decitabine 10mg/m2) | Dose Level 3 (Decitabine 15 mg/m2) | Total
Number analyzed (Participants) | 3 | 22 | 12 | 37
Age, Continuous [Median (Full Range); unit: Years] | 11.18 [2.47 to 12.83] | 7.59 [1.88 to 20.13] | 11.46 [1 to 20.51] | 8.4 [1.0 to 20.51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 3 | 12
  Male | 2 | 14 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 7
  Not Hispanic or Latino | 2 | 16 | 8 | 26
  Unknown or Not Reported | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 1 | 13 | 9 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 3 | 21 | 11 | 35
  Australia | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Dose of Decitabine That Can be Safely Given With Vorinostat, Fludarabine, High Dose Cytarabine and G-CSF (FLAG)
Description: The incidence of dose limiting toxicity (DLT) will be measured. The maximum tolerated dose will be the highest study dose at which 1 or fewer of six patients experience DLT during cycle 1 of therapy
Time Frame: during course 1 DLT evaluation period, approx 9 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: Decitabine = 7.5 mg/m2
- Dose Level 2: Decitabine = 10 mg/m2
- Dose Level 3: Decitabine = 15mg/m2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 22 | 12
Participants
  Patient completed therapy without DLT | 3 | 20 | 12
  Patient experienced DLT | 0 | 0 | 0
  Patients withdrew or not evaluable | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Through 30 days after the last day of protocol therapy (Cycle 1 only), approximately 9 weeks total duration.
Arm/Group | Dose Level 1 (Decitabine = 7.5mg/m2) | Dose Level 2 (Decitabine 10mg/m2) | Dose Level 3 (Decitabine 15 mg/m2)
All-Cause Mortality (participants affected / at risk) | 3/3 | 22/22 | 12/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 18/22 | 12/12
Other Adverse Events (participants affected / at risk) | 3/3 | 22/22 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (Decitabine = 7.5mg/m2) (N=3) | Dose Level 2 (Decitabine 10mg/m2) (N=22) | Dose Level 3 (Decitabine 15 mg/m2) (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0
Heart Failure (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Edema Limbs (General disorders) | 0 | 1 | 0
Encephalitis Infection (Infections and infestations) | 0 | 0 | 1
Disseminated Fungal Infection (Trichosporon Asahii) (Infections and infestations) | 0 | 1 | 0
Fungemia Candida Parapsilosis Blood Line Infection (Infections and infestations) | 0 | 1 | 0
Candida Parapsilosis (Infections and infestations) | 0 | 0 | 1
Disseminated Fungal, Mucor (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 3
Lung Infection (Infections and infestations) | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Infections and infestations) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Leukemia Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 0 | 1 | 0
Paraplegia NOS (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Bilateral Erythematous Knee Lesions (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (Decitabine = 7.5mg/m2) (N=3) | Dose Level 2 (Decitabine 10mg/m2) (N=22) | Dose Level 3 (Decitabine 15 mg/m2) (N=12)
Anemia (Blood and lymphatic system disorders) | 3 | 20 | 11
Positive Blood Culture (MRSE) (Blood and lymphatic system disorders) | 0 | 1 | 0
PICC Line Bleeding (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 10 | 6
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Non-specific ST and T Wave Abnormality (Cardiac disorders) | 0 | 1 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 0 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 6 | 4
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 2 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0
Itching, Burning (Eye disorders) | 0 | 0 | 1
Vision Loss (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 3 | 1
Flashing Lights (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 5 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 8 | 2
Constipation (Cardiac disorders) | 0 | 7 | 3
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 5 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gingival Erythemia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Mucositis Oral (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 9 | 7
Oral Pain (Gastrointestinal disorders) | 0 | 2 | 0
Rectal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 6 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0
Edema Face (General disorders) | 0 | 1 | 0
Facial Pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 0
Fever (General disorders) | 2 | 10 | 5
Pain (General disorders) | 1 | 3 | 1
Neck Edema (General disorders) | 0 | 1 | 0
Localized Edema - Scrotum (General disorders) | 0 | 1 | 0
Localized Edema (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 3 | 2
Allergic reaction (Immune system disorders) | 0 | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Bacteremia (Infections and infestations) | 0 | 1 | 0
Blood infection (Infections and infestations) | 0 | 0 | 1
Coagulase Negative Staphylococcus (Infections and infestations) | 0 | 0 | 1
Oral Mucosa (Infections and infestations) | 0 | 1 | 0
HHV6 (Infections and infestations) | 0 | 1 | 0
Escherichia Coli (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Alpha Streptococcus not Streptococcus Pneumoniae, Group A or B (Infections and infestations) | 0 | 0 | 1
Human Rhinovirus (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 0
Skin Infection (Infections and infestations) | 0 | 2 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 3
Lung Infection (Infections and infestations) | 1 | 4 | 3
Nail Infection (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head Bump with Small Scab (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 3 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 9 | 5
Alkaline Phosphatase Increased (Investigations) | 2 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 10 | 5
Blood Bilirubin Increased (Investigations) | 1 | 9 | 3
CD4 Lymphocytes decreased (Investigations) | 0 | 1 | 0
Creatinine Increased (Investigations) | 0 | 1 | 2
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 1 | 2 | 0
Fibrinogen Decreased (Investigations) | 0 | 1 | 0
INR Increased (Investigations) | 0 | 2 | 1
Hyperphosphatemia (Investigations) | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 14 | 8
Lymphocyte Count Increased (Investigations) | 0 | 3 | 0
Neutrophil Count Decreased (Investigations) | 3 | 19 | 7
Platelet Count Decreased (Investigations) | 3 | 19 | 11
Weight Gain (Investigations) | 0 | 2 | 0
Weight Loss (Investigations) | 1 | 5 | 2
White Blood Cell Decreased (Investigations) | 3 | 18 | 10
Ejection Fraction Decreased (Investigations) | 0 | 2 | 0
Hemoglobin Increased (Investigations) | 0 | 1 | 0
GGT Increased (Investigations) | 1 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 7 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 9 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 4 | 3
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 13 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 8 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 15 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 5 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 11 | 7
Hypophosphatemia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Physical Deconditioning (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle Weakness Trunk (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Lethargy (Nervous system disorders) | 0 | 1 | 0
Pseudotumor Cerebri (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 2
Confusion (Psychiatric disorders) | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 2 | 0
Hematuria (Renal and urinary disorders) | 0 | 3 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Urinary Tract Pain (Renal and urinary disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0
Penile Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
RSV Virus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Parainfluenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinovirus (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Pressure Injury of Buttock (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin and Subcutaneous Tissue Disorders - Other Specify: Fungal Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythematous Knee Lesion, Right Knee (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Macular Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Irritation at G Tube Site (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 7 | 4
Hypotension (Vascular disorders) | 0 | 6 | 3
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03263936/Prot_SAP_ICF_000.pdf